CLINICAL TRIAL: NCT02187848
Title: A First-in-Human Study for the Evaluation of the Safety, Pharmacokinetics and Antitumor Activity of SAR408701 in Patients With Advanced Solid Tumors
Brief Title: Evaluation of SAR408701 in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision, The decision is not related to any safety concern.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TED13751; U1111-1153-3461 (Registry Identifier: ICTRP); 2014-001130-29 (EudraCT Number)
Record Dates: First submitted 2014-06-24; First posted 2014-07-11 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms | interventions — tusamitamab ravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (9):
- SAR408701 Main Dose Escalation Cohort (Experimental): Dose escalation administered intravenously, once every two weeks
  Interventions: Drug: SAR408701
- SAR408701 Expansion Cohort colorectal cancer (CRC) (Experimental): Administered intravenously at the maximum tolerated dose (MTD), once every 2 weeks, to patients with colorectal cancer
  Interventions: Drug: SAR408701
- SAR408701 Expansion Cohort non-squamous NSCLC (Experimental): Administered intravenously at the MTD, once every 2 weeks, to patients with carcinoembryonic antigen-related cell adhesion molecule 5 (CEACAM5) expressing non-squamous non-small cell lung cancer (NSCLC) of at least 50% of tumor cells at or above 2+ intensity
  Interventions: Drug: SAR408701
- SAR408701 Expansion Cohort gastric adenocarcinoma (Experimental): Administered intravenously at the MTD, once every 2 weeks, to patients with CEACAM5 expressing gastric adenocarcinoma
  Interventions: Drug: SAR408701
- SAR408701 Loading Dose Escalation cohorts (Escalation bis) (Experimental): Loading dose escalation administered intravenously at first cycle, followed by MTD, once every 2 weeks
  Interventions: Drug: SAR408701
- SAR408701 Expansion Cohort non-squamous NSCLC (Lung bis) (Experimental): Administered intravenously at the MTD, once every 2 weeks, to patients with CEACAM5 expressing non-squamous NSCLC of at least 1% but below 50% of tumor cells at or above 2+ intensity
  Interventions: Drug: SAR408701
- SAR408701 Expansion Cohort colorectal cancer (CRC-L) (Experimental): Loading dose of determined MTD-L administered intravenously at first cycle, followed by MTD, once every 2 weeks
  Interventions: Drug: SAR408701
- SAR408701 Expansion Cohort small cell lung cancer (SCLC) (Experimental): Administered intravenously at the MTD, once every 2 weeks, to patients with CEACAM5 expressing SCLC
  Interventions: Drug: SAR408701
- SAR408701 Dose Escalation every 3 weeks cohort (Experimental): Dose escalation administered intravenously, once every three weeks
  Interventions: Drug: SAR408701

INTERVENTIONS:
Drug: SAR408701 — Pharmaceutical form: concentrate for solution for infusion Route of administration: intravenous

SUMMARY:
Primary Objectives:

* To determine the maximum tolerated dose (MTD) of SAR408701 administered as monotherapy, once every 2 weeks (with and without a loading dose at Cycle 1) to patients with advanced solid tumors (Main Escalation and Loading Dose Escalation Q2W).
* To determine the maximum tolerated dose (MTD) of SAR408701 administered as monotherapy, once every 3 weeks to patients with advanced solid tumors (Escalation Q3W Cycle).
* To assess efficacy according to Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) (Expansion Phase) when SAR408701 is administered once every 2 weeks with or without a loading dose at Cycle 1.

Secondary Objectives:

* To characterize the overall safety profile of SAR408701.
* To characterize the pharmacokinetic (PK) profile of SAR408701 and of its potential circulating derivatives.
* To identify the recommended phase 2 dose (RP2D) of SAR408701.
* To assess the potential immunogenicity of SAR408701.

DETAILED DESCRIPTION:
The study duration for an individual patient will start from the signature of the informed consent, will include a period to assess eligibility (screening period) of up to approximately 4 weeks (28 days), a treatment period and an end-of-treatment visit around 30 days following the last administration of study drug, and at least one follow-up visit after the end-of-treatment visit. Additional follow-up visits may be required until resolution or stabilization of adverse events (at least 30 days). Treatment may continue until precluded by toxicity, progression, or upon patient's request. If the patient stops study treatment for reason other than disease progression, follow-up visit will be performed every 3 months until disease progression or initiation of another anti-tumor treatment or death, whichever comes first.

ELIGIBILITY:
Inclusion criteria:

* Locally advanced or metastatic solid malignant tumor disease for which no standard alternative therapy is available.
* Availability of archived tumor tissue for carcinoembryonic antigen-related cell adhesion molecule 5 (CEACAM5 or CEA) testing.
* For participants in the Dose Escalation Cohorts (Main Escalation and Loading Dose Cohorts at every 2 week cycle and Dose Escalation every 3 week cycle): patients with tumors expressing or likely to be expressing CEACAM5 which includes colorectal cancer (CRC), non-squamous non-small cell lung cancer (NSCLC), gastric adenocarcinoma, squamous cell carcinoma of the cervix, pancreas adenocarcinoma, bladder transitional cell carcinoma, cholangiocarcinoma, epithelial ovarian cancer and endometrial adenocarcinoma are favored, or if carcinoembryonic antigen (CEA) plasma levels >5 ng/mL.
* For participants to the Expansion Phase cohorts: patients with CRC or with CEACAM5 positive non-squamous NSCLC, small cell lung cancer (SCLC) or gastric carcinoma (including esophago-gastric junction adenocarcinoma of the Siewert types II and III).
* At least one measurable lesion by RECIST v1.1 in the Expansion Phase only.
* At least one lesion amenable to biopsy (Expansion cohort - CRC and gastric cancer only). Patient must consent to a baseline biopsy for retrospective confirmation of tumor CEACAM5 expression, except if NSCLC or SCLC without lesion amenable to biopsy.
* Signed informed consent.

Exclusion criteria:

* Aged less than 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status more than 1.
* New or progressing brain involvement.
* Concurrent treatment with any other anticancer therapy or inadequate wash-out period for prior anticancer therapies before first administration of SAR408701, or non-resolution of toxicities induced by these anticancer therapies.
* Female or male patients with reproductive potential who do not agree to use an accepted effective method of contraception during the study treatment period and for at least 3 months following completion of study treatment.
* Pregnancy or breast-feeding.
* Participation to any clinical research study evaluating another investigational drug or therapy within 3 weeks of initiation of study regimen.
* Prior therapy targeting CEACAM5.
* Prior maytansinoid treatments (DM1 or DM4 antibody drug conjugates).
* Poor bone marrow reserve resulting in low blood cell counts.
* Poor kidney and liver functions.
* Any of the following within 6 months prior to study enrolment: infectious or inflammatory bowel disease, diverticulitis, gastrointestinal perforation, intestinal obstruction, and gastrointestinal hemorrhage. Patients with malabsorption syndrome are excluded.
* Previous history and or unresolved corneal disorders. The use of contact lenses is not permitted.
* Unresolved signs and symptoms of neuropathy; Grade 1 is acceptable if prior neurotoxic drugs such as cisplatin or taxanes.
* Abnormal cardiac function defined by a left ventricular ejection fraction (LVEF) of <50%.
* Cardiac conduction defects, or any other clinically significant arrhythmias.
* Known intolerance to infused protein products.
* Medical conditions requiring concomitant administration of medications with narrow therapeutic window, metabolized by cytochrome P450 (CYPs) enzymes and for which a dose reduction cannot be considered.
* Medical conditions requiring concomitant administration of strong CYP3A inhibitor, unless it can be discontinued at least 2 weeks before 1st administration of SAR408701.
* Contraindications to the use of ophthalmic vasoconstrictor and/or corticosteroid as per package insert of each drug, including the following: increase intraocular pressure, prior or current glaucoma, narrow-angle glaucoma, ongoing eye infection, uncontrolled hypertension, known/suspected allergy to constituents of the preparation (such as sodium bisulfite).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2014-07-23 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Number of dose limiting adverse events (every 2 week cycle) | 4 weeks
Assessment of overall response rate using standard imaging and RECIST 1.1 criteria | Up to 40 months
Number of dose limiting adverse events (every 3 week cycle) | 3 weeks

SECONDARY OUTCOMES:
Number of treatment emergent adverse events | Up to 4 years
Maximum concentration (Cmax) | 2 months
Time to reach maximum concentration (tmax) | 2 months
Trough plasma concentrations (Ctrough) | Intensive testing within first 2 months, then every 2 weeks
Area under the plasma concentration versus time curve between 0 and 14 days (AUC0-14day) for Q2W or between 0 and 21 days (AUC-21 day) for Q3W | 2 months
Mean systemic clearance (CL) | 2 months
Clearance at steady state (CLss) | 2 months
Accumulation ratio (Rac) on AUC0-14day and Cmax | 2 months
Detection of the development of anti-SAR408701 antibody | Up to 40 months
Duration of response | Up to 40 months - assessment every 6-8 weeks
Time to Progression | Up to 40 months - assessment every 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (20):
- United States (2):
  - Yale University School of Medicine Site Number : 840002, New Haven, Connecticut
  - Dana Farber Cancer Institute- Site Number : 840005, Boston, Massachusetts
- Investigational Site Number : 124001, Toronto, Ontario, Canada
- France (7):
  - Investigational Site Number : 250003, Bordeaux
  - Investigational Site Number : 250006, Dijon
  - Investigational Site Number : 250004, Marseille
  - Investigational Site Number : 250007, Rennes
  - Investigational Site Number : 250005, Saint-Mandé
  - Investigational Site Number : 250002, Toulouse
  - Investigational Site Number : 250001, Villejuif
- South Korea (5):
  - Investigational Site Number : 410002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 410005, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 410003, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 410004, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 410001, Seoul, Seoul-teukbyeolsi
- Spain (5):
  - Investigational Site Number : 724001, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 724002, Majadahonda, Madrid
  - Investigational Site Number : 724003, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 724004, Madrid / Madrid, Madrid, Comunidad de
  - Investigational Site Number : 724006, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Gazzah A, Bedard PL, Hierro C, Kang YK, Abdul Razak A, Ryu MH, Demers B, Fagniez N, Henry C, Hospitel M, Soria JC, Tabernero J. Safety, pharmacokinetics, and antitumor activity of the anti-CEACAM5-DM4 antibody-drug conjugate tusamitamab ravtansine (SAR408701) in patients with advanced solid tumors: first-in-human dose-escalation study. Ann Oncol. 2022 Apr;33(4):416-425. doi: 10.1016/j.annonc.2021.12.012. Epub 2022 Jan 10. PMID 35026412
- [Result] Tabernero J, Bedard PL, Bang YJ, Vieito M, Ryu MH, Fagniez N, Chadjaa M, Soufflet C, Masson N, Gazzah A. Tusamitamab Ravtansine in Patients with Advanced Solid Tumors: Phase I Study of Safety, Pharmacokinetics, and Antitumor Activity Using Alternative Dosing Regimens. Cancer Res Commun. 2023 Aug 28;3(8):1662-1671. doi: 10.1158/2767-9764.CRC-23-0284. eCollection 2023 Aug. PMID 37645622
- [Derived] Gazzah A, Ternes N, Lee JS, Wang E, Carene D, Wang H, Masson N, Boitier E, Lartigau A, Mace N, Chadjaa M, Dib C, Nunes M, Muzard G, Longuemaux-Valence S, Bauchet AL. Biomarker analysis from a Phase 1/1b study of tusamitamab ravtansine in patients with advanced non-small cell lung cancer. Transl Oncol. 2026 Jan;63:102615. doi: 10.1016/j.tranon.2025.102615. Epub 2025 Dec 3. PMID 41337813